CLINICAL TRIAL: NCT06945783
Title: A Randomized Controlled Trial on the Effect of Kinesio Taping on Balance and Functionality in Patients With Nonspecific Low Back Pain
Brief Title: Kinesio Taping for Balance and Function in Low Back Pain
Acronym: KTFB-NSLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Dilara Durmaz (Other)
Responsible Party: Sponsor-Investigator, Elif Dilara Durmaz, invenstigator, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ISU_NSLBP_KT_2025
Record Dates: First submitted 2025-03-19; First posted 2025-04-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Balance Disorders; Low Back Pain
Keywords: Kinesiology Taping; Nonspecific Low Back Pain; Physiotherapy
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Model Description:
  Participants were assigned to either an intervention group receiving kinesiology taping combined with physiotherapy or a control group receiving physiotherapy alone. Both groups were treated in parallel and assessed pre- and post-intervention.
Masking Description: No masking was applied. Both participants and investigators were aware of the assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesiology Taping + Physiotherapy (Experimental): Participants in this group received kinesiology taping applied to the lumbar region in addition to a physiotherapy program that included therapeutic exercises and modalities tailored for nonspecific low back pain. The intervention aimed to improve balance, reduce pain, and enhance functional outcomes.
  Interventions: Device: Kinesiology Taping; Other: Physiotherapy
- Physiotherapy Only (Active Comparator): Participants in this group received only the physiotherapy program, which included therapeutic exercises and modalities commonly used in the treatment of nonspecific low back pain. No kinesiology taping was applied in this group.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: Kinesiology Taping — Kinesiology taping was applied to the lumbar area of the participants in the intervention group. The taping aimed to improve posture, reduce pain, and enhance balance and functional performance.
  Arms: Kinesiology Taping + Physiotherapy
Other: Physiotherapy — The physiotherapy program included therapeutic exercises and physical modalities (such as stretching, strengthening, and posture training) tailored for individuals with nonspecific low back pain.

SUMMARY:
This study aims to examine the effects of kinesiology taping on balance and functional ability in individuals with nonspecific low back pain. Nonspecific low back pain is a common condition that is not linked to a specific medical cause and is often associated with balance problems, reduced physical function, and psychological challenges. In this study, 35 patients aged between 18 and 65 were included. One group received kinesiology taping along with physiotherapy, while the other group received only physiotherapy.

DETAILED DESCRIPTION:
Nonspecific low back pain (NSLBP) is a common musculoskeletal condition that cannot be attributed to a specific pathology. It often leads to limitations in functional activities, impaired balance, and psychological distress, such as depressive symptoms. This study investigates the effects of kinesiology taping on balance and functional outcomes in individuals diagnosed with NSLBP.

The study was conducted on 35 participants aged 18 to 65 years. Participants were randomly assigned to two groups: the intervention group received kinesiology taping in combination with physiotherapy, while the control group received only physiotherapy treatment. Various outcome measures were used to assess the effects of the interventions, including the Visual Analog Scale (VAS) for pain intensity, Functional Rating Index (FRI), Modified Oswestry Disability Index (MODI), Beck Depression Inventory (BDI), Nottingham Health Profile (NHP), and the Flamingo Balance Test.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* Diagnosis of nonspecific low back pain
* Duration of low back pain longer than 6 weeks
* Ability to attend an outpatient physiotherapy program

Exclusion Criteria:

* History of spinal surgery
* Presence of neurological deficits on physical examination
* Contraindication to kinesiology taping
* Pregnancy
* Cardiovascular or pulmonary diseases that contraindicate exercise
* History of lower extremity surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Functional Rating Index (FRI) score | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Functional status was assessed using the Functional Rating Index (FRI) to evaluate the level of functional disability related to nonspecific low back pain. A decrease in the score indicates improved functional status.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) score for pain | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Pain intensity was evaluated using the Visual Analog Scale. A decrease in score indicates reduced pain severity.
Change in Flamingo Balance Test (FBT) score | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Balance was assessed using the Flamingo Balance Test. Improved performance indicates better postural control and balance.
Change in Beck Depression Inventory (BDI) score | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Psychological status was assessed using the Beck Depression Inventory. A decrease in score reflects improved mood and reduced depressive symptoms.
Change in Oswestry Disability Index (ODI) score | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Disability level related to low back pain was evaluated using the Oswestry Disability Index. A decrease in score reflects improved functional ability.
Change in Nottingham Health Profile (NHP) score | Baseline (Day 1)": Initial assessment (Day 1 of the study) "3 weeks post-intervention": Second assessment, 3 weeks after the intervention (after the treatment program)
  Health-related quality of life was evaluated using the Nottingham Health Profile. A decrease in score indicates better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Universyt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes